CLINICAL TRIAL: NCT05235256
Title: Lecturer of Anesthesia- Anesthesia Department Ain Shams University
Brief Title: Sphenopalatine Block Versus Greater Occipital Nerve Block in PDPH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU R 80/2021
Record Dates: First submitted 2021-11-16; First posted 2022-02-11 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Lidocaine; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPGB Group (Active Comparator): patients will receive bilateral sphenopalatine ganglion block using 3ml mixture of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each nostril).
  Interventions: Procedure: bilateral sphenopalatine ganglion block; Drug: lidocaine plus dexamethasone
- GONB Group (Active Comparator): patients will receive bilateral greater occipital nerve block using a mixture of 3ml of 2ml 2% lidocaine plus 1ml dexamethasone 4mg (on each side of the occipital region).
  Interventions: Procedure: bilateral greater occipital nerve block; Drug: lidocaine plus dexamethasone

INTERVENTIONS:
Procedure: bilateral sphenopalatine ganglion block — peripheral n block
  Arms: SPGB Group
Procedure: bilateral greater occipital nerve block — bilateral greater occipital nerve block
  Arms: GONB Group
Drug: lidocaine plus dexamethasone — lidocaine plus dexamethasone

SUMMARY:
Management of postdural puncture headache (PDPH) has always been challenging for anesthesiologists. PDPH not only increases the misery of the patient, but the length of stay and overall cost of treatment in the hospital also increases. Although the epidural blood patch ( EBP ) is an effective way of treating the problem, the procedure itself could cause another inadvertent dural puncture (DP). Moreover, sometimes patients need to have a second EBP, if the first one is not completely effective. This can be difficult to explain to the patient who has already suffered a lot. Peripheral nerve blocks are well tolerated and effective as adjunctive therapy for many disabling headache disorder.

Sphenopalatine ganglion is a parasympathetic ganglion, located in the pterygopalatine fossa. Transnasal sphenopalatine ganglion block ( SPGB ) has been successfully used to treat chronic conditions such as migraine, cluster headache, and trigeminal neuralgia, and may be a safer alternative to treat PDPH: It is minimally invasive and carried out at the bedside without using imaging. Besides that, it has apparently a faster start than EBP, with better safety profile.

Another minimally invasive peripheral nerve block which has been used quite successful is greater occipital nerve block (GONB). The GONB has been in use for more than a decade to treat complex headache syndromes of varying etiologies like migraine , cluster headache and chronic daily headache with encouraging results. Greater Occipital Nerve (GON) arises from C2-3 segments, its most proximal part lies between obliqua capitis inferior and semispinalis, near the spinous process. Then, GON enters into semispinalis passing through it and after its exit; it enters into trapezius muscle. In distal region of trapezius fascia, it is crossed by the occipital artery and finally the nerve exits the trapezius fascia insertion into the nuchal line about 5-cm lateral to midline. Functionally, GON supplies major rectus capitis posterior muscle, and the skin, muscles, and vessels of the scalp, but is the main sensory supply of occipital region.

Many providers believe that the local anesthetic produces the rapid onset of headache relief, like an abortive agent, and that the locally acting steroid produces the preventive like action of up to 6 weeks as dexamethasone possess potent anti inflammatory and immunosuppressive actions by inhibiting cytokine-mediated pathways .

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients ( American Society of Anesthesiologists ) ASA I&II ,body weight between 60-100kg expressing PDPH after spinal anesthesia, (VAS > 4 ) with standard treatment such as intravenous fluids, abdominal binder, bed rest and caffeine.

Exclusion Criteria:

* • ASA III& IV patients.

  * Refusal of the patient.
  * Patients with chronic headache or migraine.
  * Hypertensive patients.
  * A patient that cannot comply with the VAS.
  * Infection at site of the block
  * Known coagulation defect.
  * Nasal septal deviation, polyp, history of nasal bleeding.
  * Allergy to local anaesthetics.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS ) | first 24 hours after the procedure
  Visual A nalogue Scale will be used to asses the efficacy of either SPGB or GONB for treatment of PDPH .Score from 0 to 100 (0=no pain, 100=most severe pain)

SECONDARY OUTCOMES:
total analgesic consumption | first 24 hours after the block
  total dose of ketorolac will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt